CLINICAL TRIAL: NCT06540586
Title: Evaluation of the Postoperative Analgesic Efficacy of Modified Thoracoabdominal Plane Block With Perichondral Approach and Quadratus Lumborum Block in Laparoscopic Cholecystectomies
Brief Title: Postoperative Analgesic Efficacy of Modified TAPA and QL Blocks in Laparoscopic Cholecystectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, SERPİL ŞEHİRLİOĞLU, MD, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GaziosmanpasaTREHTA
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pain Management; Postoperative Pain; Analgesia; Nerve Blocks; Cholecystectomy
Keywords: postoperative pain; laparoscopic cholecystectomy; quadratus lumborum block; m-tapa block; abdominal wall blocks; postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quadratus lumborum block group (Active Comparator): Patients are placed in the lateral decubitus position. The area where the block will be applied is disinfected with povidine iodine. A convex ultrasound probe is placed on the midaxillary line above the iliac crest. By visualizing the transverse process adjacent to the psoas major and quadratus lumborum muscles, using the in-plane technique, using a 22 gauge 80 mm peripheral block needle after negative aspiration into the anterior layer of the thoracolumbar fascia anterior to the quadratus lumborum muscle muscle, 0.5-1 ml of serum After observing hydrodissection with physiological, 20 ml of 0.25% bupivacaine is injected. The same is done to the opposite side.
  Interventions: Procedure: anterior Quadratus lumborum block
- m-tapa block (Active Comparator): In the M-TAPA block group, with the patient in the supine position, a linear high-frequency linear ultrasound (USG) probe is angled to visualize the inferior surface of the costochondral junction at the level of the 10th costochondral cartilage. Under sterile conditions, using the in-plane technique with a 22G 80 mm peripheral block needle, the needle is advanced posterior to the 10th costal cartilage by taking the lower edge of the cartilage in the sagittal plane as the midline. After hydrodissection with 2-3 ml isotonic saline to confirm the site, 20 ml of 0.25% Bupivacaine is administered under USG guidance. The same procedure is performed on the contralateral side as well.
  Interventions: Procedure: M-TAPA BLOCK

INTERVENTIONS:
Procedure: anterior Quadratus lumborum block — Patients are placed in the lateral decubitus position. The area where the block will be applied is disinfected with povidine iodine. A convex ultrasound probe is placed on the midaxillary line above the iliac crest. By visualizing the transverse process adjacent to the psoas major and quadratus lumborum muscles, using the in-plane technique, using a 22 gauge 80 mm peripheral block needle after negative aspiration into the anterior layer of the thoracolumbar fascia anterior to the quadratus lumborum muscle muscle, 0.5-1 ml of serum After observing hydrodissection with physiological, 20 ml of 0.25% bupivacaine is injected. The same is done to the opposite side.
  Arms: Quadratus lumborum block group
Procedure: M-TAPA BLOCK — In the M-TAPA block group, with the patient in the supine position, a linear high-frequency linear ultrasound (USG) probe is angled to visualize the inferior surface of the costochondral junction at the level of the 10th costochondral cartilage. Under sterile conditions, using the in-plane technique with a 22G 80 mm peripheral block needle, the needle is advanced posterior to the 10th costal cartilage by taking the lower edge of the cartilage in the sagittal plane as the midline. After hydrodissection with 2-3 ml isotonic saline to confirm the site, 20 ml of 0.25% Bupivacaine is administered under USG guidance. The same procedure is performed on the contralateral side as well.
  Arms: m-tapa block

SUMMARY:
Comparison of Postoperative Analgesic Effects of M-TAPA and Anterior Quadratus Lumborum Blocks in Laparoscopic Cholecystectomies.

DETAILED DESCRIPTION:
In trunk blocks, the interfascial area between the anterior abdominal wall or back muscles is targeted. Local anesthetics are used for this purpose. Since there is no blood circulation and vascularization in the interfascial areas, the absorption of local anesthetics is slow, providing long-lasting analgesia. Therefore, they are used as a part of multimodal analgesia. The effectiveness of trunk blocks can vary depending on the patient's anatomical differences and previous surgeries, but on average, analgesic effectiveness lasts for 8-12 hours. Sometimes analgesic effectiveness extending up to 24 hours has been reported.

In laparoscopic cholecystectomy operations, pain plays a role in postoperative atelectasis, pneumonia due to atelectasis, prolonged hospital stay, and discharge. To reduce the use of opioids due to their side effects such as nausea, vomiting, itching, constipation, and addiction, opioid-free analgesia is applied, and regional techniques are used. Quadratus lumborum blocks and M-TAPA blocks have been safely and easily applied in abdominal surgery in recent years thanks to developments in trunk blocks and ultrasound technology, and they are frequently preferred.

ELIGIBILITY:
* Inclusion Criteria:
* scheduled for elective Laparoscopic chplecystectomy
* Patients aged ≥18 years
* American Society of Anesthesiologists physical status (ASA) Ⅰ-II

Exclusion Criteria:

ASA III-IV patient

* local anesthetic allergy
* Infection at the procedure site Body Mass Index >35 kg/m2 Anticoagulant use with bleeding disorder Chronic analgesia and opioid use with mental and psychiatric disorders Contraindications to regional anesthesia several lung and heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Total amount of opioid requirements | within 24 hours after the surgery
  The total tramadol use of the patients in 24 hours will be recorded.

SECONDARY OUTCOMES:
rescue analgesia | within 24 hours after the surgery
  The rescue analgesia requirement and time of the need of the rescue analgesia requirement

OTHER OUTCOMES:
intraoperative remifentanil consumption | during operation procedure]
  The total remifentanil use to be used in the maintenance of 0.05-0.2 mcg/kg remifentanil will be recorded by titration according to the hemodynamic data of the intraoperative patients.
Visual Analogue Scale values | at 1st, 4th,8th 12th and 24th hours after the surgery]
  Visual Analogue Scale is a scale of 0-10 cm in length, expressed by non-standard verbal descriptors (no pain-unbearable pain..) indicating the limits of pain intensity on both sides, horizontally or vertically.
side effects such as nausea, vomiting and shoulder pain | within 24 hours after the surgery
  The incidence of postoperative side effects such as nausea, vomiting and shoulder pain will be evaluated.a

CONTACTS AND LOCATIONS:
Overall Officials: serpil sehirlioglu, MD, Principal Investigator — Gaziosmanpasa Research and Education Hospital; turan aydemir, MD, Study Director — Gaziosmanpasa Research and Education Hospital; döndü moralar, MD, Study Director — Gaziosmanpasa Research and Education Hospital
Locations (1):
- Gaziosmanpasa Research and Education Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elsharkawy H, El-Boghdadly K, Barrington M. Quadratus Lumborum Block: Anatomical Concepts, Mechanisms, and Techniques. Anesthesiology. 2019 Feb;130(2):322-335. doi: 10.1097/ALN.0000000000002524. No abstract available. PMID 30688787
- [Background] Aygun H, Kavrut Ozturk N, Pamukcu AS, Inal A, Kiziloglu I, Thomas DT, Tulgar S, Nart A. Comparison of ultrasound guided Erector Spinae Plane Block and quadratus lumborum block for postoperative analgesia in laparoscopic cholecystectomy patients; a prospective randomized study. J Clin Anesth. 2020 Jun;62:109696. doi: 10.1016/j.jclinane.2019.109696. Epub 2019 Dec 18. PMID 31862217
- [Background] Tulgar S, Selvi O, Thomas DT, Deveci U, Ozer Z. Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) provides effective analgesia in abdominal surgery and is a choice for opioid sparing anesthesia. J Clin Anesth. 2019 Aug;55:109. doi: 10.1016/j.jclinane.2019.01.003. Epub 2019 Jan 9. No abstract available. PMID 30639940